CLINICAL TRIAL: NCT00758498
Title: A 3-Day, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of the Effect of Armodafinil Treatment (50 and 150 mg/Day) in Healthy Subjects With Excessive Sleepiness Associated With Jet Lag Disorder
Brief Title: Study of the Effect of Armodafinil Treatment in Healthy Subjects With Excessive Sleepiness Associated With Jet Lag Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C10953/3065/ES/MN
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2010-07-08 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Excessive Sleepiness
MeSH Terms: conditions — Disorders of Excessive Somnolence | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): armodafinil - dosage of 50 mg/day
  Interventions: Drug: armodafinil
- 2 (Experimental): armodafinil - dosage of 150 mg/day
  Interventions: Drug: armodafinil
- 3 (Placebo Comparator): matching placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: armodafinil — 50 mg/day orally, once daily in the morning for 3 days
  Arms: 1
Drug: armodafinil — 150 mg/day orally, once daily in the morning for 3 days
  Arms: 2
Drug: placebo — placebo tablets, once daily in the morning for 3 days
  Arms: 3

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group study of armodafinil and placebo treatment in healthy subjects with excessive sleepiness associated with jet lag disorder.

ELIGIBILITY:
Key Inclusion Criteria:

* History of jet lag symptoms during the past 5 years.
* The subject is in good health, as determined by a medical and psychiatric history, medical examination, clinical laboratory test results, and electrocardiography (ECG) and physical examination findings.
* Women of childbearing potential must be abstinent or use a medically accepted method of contraception, and must continue use of this method for the duration of the study (and for 30 days after participation in the study).
* The subject is willing to comply with study restrictions and remain at the study center overnight, as required.
* The subject must agree to refrain from alcohol use during the study.
* The subject has a valid U.S. passport

Key Exclusion Criteria:

* The subject has a history (past 12 months) or diagnosis of narcolepsy, obstructive sleep apnea/hypopnea syndrome (OSAHS), shift work sleep disorder (SWSD), or any other sleep disorder associated with excessive daytime sleepiness; or the subject has a history or current diagnosis of hypersomnia, insomnia, or sleep disorder.
* The subject has any serious acute or chronic cardiovascular, pulmonary, gastrointestinal, neurological, endocrine or renal illness (including diabetes mellitus), hepatitis, asthma, chronic obstructive pulmonary disease (COPD), or any other clinically relevant significant medical condition.
* The subject has a history of any cutaneous drug reaction or drug hypersensitivity, or any clinically significant hypersensitivity reaction, or multiple allergies.
* The subject has a history of deep vein thrombosis (DVT).
* The subject has known human immunodeficiency virus (HIV).
* The subject is pregnant or lactating.
* The subject has used nicotine within the last 3 months.
* The subject has a history of seizures, except for a single febrile seizure.
* The subject has a psychiatric disorder that would affect participation in the study or full compliance with study procedures.
* The subject has a clinically significant deviation from normal in clinical laboratory results, vital signs measurements, or physical examination findings.
* The subject used any prescription or over the counter drugs disallowed by the protocol within 7 days of screening visit 2 (i.e., stimulants, hypnotics).
* The subject has used an investigational drug within 1 month before the screening visit.
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion.
* The subject has a known hypersensitivity to armodafinil or modafinil, or any other component of the study drug tablets.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon
Locations (4):
- United States (4):
  - Neurotrials Research, Inc., Atlanta, Georgia
  - Community Research, Crestview, Kentucky
  - Clinilabs, Inc., New York, New York
  - SleepMed of South Carolina, Columbia, South Carolina

REFERENCES:
- [Derived] Rosenberg RP, Bogan RK, Tiller JM, Yang R, Youakim JM, Earl CQ, Roth T. A phase 3, double-blind, randomized, placebo-controlled study of armodafinil for excessive sleepiness associated with jet lag disorder. Mayo Clin Proc. 2010 Jul;85(7):630-8. doi: 10.4065/mcp.2009.0778. Epub 2010 Jun 7. PMID 20530317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 centers in the United States (US; origination study centers) and 3 centers in France (destination study centers). First participant enrolled: September 2008 / Last participant last visit: February 2009
Pre-assignment Details: Study consisted of a 1 to 8 week screening period, a 3-day double blind treatment period, and a 7-day follow-up period. 1298 subjects were screened, 431 subjects met entry criteria in the US; 4 subjects were ineligible upon arrival in France (due to AEs), and 1 subject randomized to placebo did not have any post-baseline efficacy assessments.
Groups:
- Armodafinil 50 mg/Day: Subjects were randomly assigned to one of three treatment groups 1:1:1. Armodafinil 50 mg was administered orally once daily at approximately 0800 (8:00am) on days 1, 2, and 3.
- Armodafinil 150 mg/Day: Subjects were randomly assigned to one of three treatment groups 1:1:1. Armodafinil 150 mg was administered orally once daily at approximately 0800 (8:00am) on days 1, 2, and 3.
- Placebo: Subjects were randomly assigned to one of three treatment groups 1:1:1. Placebo was administered orally once daily at approximately 0800 (8:00am) on days 1, 2, and 3.
Period: Overall Study
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Started | 142 | 143 | 142
Completed | 139 | 141 | 137
Not Completed | 3 | 2 | 5
Not completed — Adverse Event | 2 | 2 | 3
Not completed — Subject legally detained out of state | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Noncompliance to study procedures | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo | Total
Number analyzed (Participants) | 142 | 143 | 142 | 427
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 142 | 143 | 142 | 427
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.7 (12.01) | 34.6 (10.38) | 36.0 (10.06) | 35.8 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 84 | 67 | 229
  Male | 64 | 59 | 75 | 198
Region of Enrollment [Number; unit: participants]
  United States | 142 | 143 | 142 | 427

OUTCOME MEASURES:

1. Primary Outcome: Mean Sleep Latency (Minutes) From the Multiple Sleep Latency Test (MSLT)- Average of Four Scheduled Naps Across Days 1 and 2
Description: MSLT is an assessment that measures likelihood of falling asleep. Mean Sleep Latency measures the time to fall asleep. On Treatment Days 1 and 2 the subject was instructed on 4 occasions to attempt to fall asleep. Each MSLT nap continued until 3 consecutive 30-second epochs of stage 1 sleep were reached, or any 30 second epoch of stage 2, 3, 4 or rapid eye movement sleep was reached. Each nap was terminated after 20 minutes if no sleep occured. Average sleep latency for the 4 naps was tabulated across days 1 and 2. Sleep latency was measured from lights out to first epoch scored as sleep.
Time Frame: Days 1 and 2
Population: Full analysis set defined as all subjects who received at least one dose of study drug and had at least one post-baseline efficacy measurement
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 142 | 143 | 141
Minutes | 7.7 (0.29) | 11.7 (0.29) | 4.8 (0.29)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Treatment was a factor and baseline value was a co-variate; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [2.07 to 3.71]
Statistical Analysis 2: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Treatment was a factor and baseline value was a co-variate; Mean Difference (Final Values) = 6.9, 95% CI 2-sided [6.06 to 7.69]

2. Primary Outcome: Average of Patient Global Impression of Severity (PGI-S) of General Condition Ratings Across Days 1 and 2
Description: The PGI-S rating scale is the patient's assessment of their general condition. The subject rates their overall condition according to the 7 following categories: 1=normal (no sign of illness), 2=borderline ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, and 7=among the most extremely ill. The term "ill" refers here to any symptoms of jet lag and overall feeling. Symptoms may include sleepiness, irritability, malaise, gastrointestinal disturbance, and level of performance. The average of PGI-S ratings across days 1 and 2 are presented here.
Time Frame: Days 1 and 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 142 | 143 | 141
Units on a scale | 1.9 (0.08) | 1.6 (0.08) | 1.9 (0.08)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.8341, ANOVA; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.20 to 0.25]
Statistical Analysis 2: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0441, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.50 to -0.05]

3. Secondary Outcome: Average of Scores Across Days 1 and 2 in the Karolinska Sleepiness Scale (KSS)
Description: The Karolinska Sleepiness Scale is a validated subject-rated instrument for measuring sleepiness, based on a scale from 1 to 9 (with 1 indicating very alert and 9 indicating very sleepy, great effort to stay awake, fighting sleep).
  The KSS was administered 5 times during the day; before each MSLT nap and before bedtime. The KSS least squares mean score across days 1 and 2 are reported here.
Time Frame: Days 1 and 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 142 | 143 | 141
Units on a scale | 4.8 (0.12) | 4.3 (0.12) | 5.5 (0.12)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA

4. Secondary Outcome: Mean Scores From the Karolinska Sleepiness Scale (KSS) at Day 1
Description: The Karolinska Sleepiness Scale is a validated subject-rated instrument for measuring sleepiness, based on a scale from 1 to 9 (with 1 indicating very alert and 9 indicating very sleepy, great effort to stay awake, fighting sleep).
  The KSS was administered 5 times during the day; before each MSLT nap and before bedtime. The KSS least squares mean score across day 1 is reported here.
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 142 | 143 | 141
Units on a scale | 5.7 (0.14) | 4.8 (0.14) | 6.3 (0.14)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0012, ANCOVA; Treatment comparisons made use of an analysis of covariance (ANCOVA) analysis with treatment as a factor and baseline value as a covariate
Statistical Analysis 2: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis by ANCOVA with treatment as a factor and the baseline value as a covariate

5. Secondary Outcome: Mean Scores From the Karolinska Sleepiness Scale (KSS) at Day 2
Description: The Karolinska Sleepiness Scale is a validated subject-rated instrument for measuring sleepiness, based on a scale from 1 to 9 (with 1 indicating very alert and 9 indicating very sleepy, great effort to stay awake, fighting sleep).
  The KSS was administered 5 times during the day; before each MSLT nap and before bedtime. The KSS Least squares mean score as measured on day 2 is reported here.
Time Frame: Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 141 | 141 | 138
Units on a scale | 4.0 (0.12) | 3.8 (0.12) | 4.7 (0.12)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Analysis of treatment comparisons is based on an analysis of variance (ANCOVA) with treatment as a factor and the baseline value as covariate
Statistical Analysis 2: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis of treatment comparisons is based on an ANCOVA with treatment as a factor and baseline value as a covariate

6. Secondary Outcome: Mean Scores From the Karolinska Sleepiness Scale (KSS) at Day 3
Description: The Karolinska Sleepiness Scale is a validated subject-rated instrument for measuring sleepiness, based on a scale from 1 to 9 (with 1 indicating very alert and 9 indicating very sleepy, great effort to stay awake, fighting sleep).
  The KSS was administered 5 times during the day; before each MSLT nap and before bedtime. The KSS least squares mean score as measured on day 3 is reported here.
Time Frame: Day 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 140 | 141 | 138
Units on a scale | 3.6 (0.10) | 3.6 (0.10) | 4.0 (0.10)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0022, ANCOVA; Analysis of treatment comparisons is based on analysis of covariance (ANCOVA) with treatment as a factor and baseline value as a covariate
Statistical Analysis 2: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0033, ANCOVA; Analysis of treatment comparisons was based on ANCOVA with treatment as a factor and the baseline as a covariate

7. Secondary Outcome: Mean Scores From the Karolinska Sleepiness Scale (KSS) Collected at Bedtime at Baseline
Description: The Karolinska Sleepiness Scale is a validated subject-rated instrument for measuring sleepiness, based on a scale from 1 to 9 (with 1 indicating very alert and 9 indicating very sleepy, great effort to stay awake, fighting sleep).
  The KSS was administered 5 times during the day; before each MSLT nap and before bedtime. The KSS mean score as measured at Baseline, collected at bedtime, is reported here.
Time Frame: Baseline prior to starting study medication
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 142 | 143 | 141
Units on a scale | 4.0 (1.71) | 4.0 (1.84) | 3.8 (1.76)

8. Secondary Outcome: Mean Scores From the Karolinska Sleepiness Scale (KSS) Collected at Bedtime at Day 1
Description: The Karolinska Sleepiness Scale is a validated subject-rated instrument for measuring sleepiness, based on a scale from 1 to 9 (with 1 indicating very alert and 9 indicating very sleepy, great effort to stay awake, fighting sleep).
  The KSS was administered 5 times during the day; before each MSLT nap and before bedtime. The KSS mean score as measured on day 1, collected only at bedtime, is reported here.
Time Frame: Day 1 bedtime
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 142 | 141 | 140
Units on a scale | 7.2 (1.97) | 6.9 (2.05) | 7.1 (2.19)

9. Secondary Outcome: Mean Scores From the Karolinska Sleepiness Scale (KSS) Collected at Bedtime at Day 2
Description: The Karolinska Sleepiness Scale is a validated subject-rated instrument for measuring sleepiness, based on a scale from 1 to 9 (with 1 indicating very alert and 9 indicating very sleepy, great effort to stay awake, fighting sleep).
  The KSS was administered 5 times during the day; before each MSLT nap and before bedtime. The KSS mean score as measured on day 2, collected only at bedtime, is reported here.
Time Frame: Day 2 bedtime
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 141 | 141 | 139
Units on a scale | 5.2 (1.96) | 5.2 (2.01) | 5.0 (2.13)

10. Secondary Outcome: Mean Scores From the Karolinska Sleepiness Scale (KSS) Collected at Bedtime at Day 3
Description: The Karolinska Sleepiness Scale is a validated subject-rated instrument for measuring sleepiness, based on a scale from 1 to 9 (with 1 indicating very alert and 9 indicating very sleepy, great effort to stay awake, fighting sleep).
  The KSS was administered 5 times during the day; before each MSLT nap and before bedtime. The KSS mean score as measured on day 3, collected only at bedtime, is reported here.
Time Frame: Day 3 bedtime
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 140 | 141 | 138
Units on a scale | 3.6 (1.71) | 3.9 (1.88) | 3.5 (1.90)

11. Secondary Outcome: Mean Ratings From the Mean Sleep Latency of the Multiple Sleep Latency Tests (MSLT) at Baseline
Description: MSLT measures the likelihood of falling asleep. Mean Sleep Latency measures the time to fall asleep (in minutes). On Treatment Days 1 and 2 the subject was instructed on 4 occasions to attempt to fall asleep. Each MSLT nap continued until 3 consecutive 30-sec epochs of stage 1 sleep were reached, or any 30 sec epoch of stage 2, 3, 4 or rapid eye movement sleep was reached. Each nap was terminated after 20 min if no sleep occurred. Sleep latency was measured from lights out to first epoch scored as sleep. Mean sleep latency from the MSLT at Baseline (Screening Day 2) is presented here.
Time Frame: Baseline defined as Screening Visit 2 within 8 weeks prior to Treatment Day 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 142 | 143 | 141
Minutes | 15.2 (3.82) | 15.3 (3.83) | 15.0 (4.17)

12. Secondary Outcome: Mean Sleep Latency (Minutes) From the Multiple Sleep Latency Tests (MSLT) at Day 1
Description: MSLT measures likelihood of falling asleep. Mean Sleep Latency measures the time to fall asleep (in minutes). On Treatment Days 1 and 2 the subject was instructed on 4 occasions to attempt to fall asleep. Each MSLT nap continued until 3 consecutive 30-sec epochs of stage 1 sleep were reached, or any 30 sec epoch of stage 2, 3, 4 or rapid eye movement sleep was reached. Each nap was terminated after 20 min if no sleep occurred. Sleep latency was measured from lights out to first epoch scored as sleep. Least squares mean sleep latency from the MSLT at day 1 is presented here.
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 142 | 143 | 141
Minutes | 5.6 (0.32) | 9.6 (0.32) | 3.4 (0.32)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis of treatment comparisons is based on analysis of covariance (ANCOVA) with treatment as factor and baseline value as a covariate
Statistical Analysis 2: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis of treatment comparisons is based on ANCOVA with treatment as factor and baseline value as a covariate

13. Secondary Outcome: Mean Sleep Latency (Minutes) From the Multiple Sleep Latency Tests (MSLT) at Day 2
Description: MSLT measures likelihood of falling asleep. Mean Sleep Latency measures the time to fall asleep (in minutes). On Treatment Days 1 and 2 the subject was instructed on 4 occasions to attempt to fall asleep. Each MSLT nap continued until 3 consecutive 30-sec epochs of stage 1 sleep were reached, or any 30 sec epoch of stage 2, 3, 4 or rapid eye movement sleep was reached. Each nap was terminated after 20 min if no sleep occurred. Sleep latency was measured from lights out to first epoch scored as sleep. Least Squares Mean sleep latency from the MSLT at day 2 is presented here.
Time Frame: Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 141 | 141 | 138
Minutes | 9.9 (0.36) | 13.8 (0.36) | 6.2 (0.36)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis of treatment comparisons is based on ANCOVA with treatment as a factor and the baseline value as a covariate; Least square mean

14. Secondary Outcome: Mean Sleep Latency (Minutes) From the Multiple Sleep Latency Tests (MSLT) at Day 3
Description: MSLT measures likelihood of falling asleep. Mean Sleep Latency measures the time to fall asleep (in minutes). On Treatment Days 1 and 2 the subject was instructed on 4 occasions to attempt to fall asleep. Each MSLT nap continued until 3 consecutive 30-sec epochs of stage 1 sleep were reached, or any 30 sec epoch of stage 2, 3, 4 or rapid eye movement sleep was reached. Each nap was terminated after 20 min if no sleep occurred. Sleep latency was measured from lights out to first epoch scored as sleep. Least Squares Mean sleep latency from the MSLT at day 3 is presented here.
Time Frame: Day 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 140 | 141 | 138
Minutes | 12.1 (0.38) | 14.8 (0.38) | 8.3 (0.39)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis of treatment comparisons are from an analysis of covariance (ANCOVA) with treatment as a factor and the baseline value as a covariate
Statistical Analysis 2: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis of treatment comparisons is from an ANCOVA with treatment as a factor and the baseline value as a covariate

15. Secondary Outcome: Mean Patient Global Impression of Severity of General Condition Ratings at Baseline
Description: The PGI-S rating scale is the patient's assessment of general condition. The subject rates their overall condition according to the 7 following categories: 1=normal (no sign of illness), 2=borderline ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, and 7=among the most extremely ill. The term "ill" refers to symptoms of jet lag including excessive sleepiness, irritability, malaise, gastrointestinal disturbance, and poor performance. The least squares mean of PGI-S ratings at Baseline is presented here.
Time Frame: Baseline, prior to start of study drug dosing
Population: Full analysis set defined as all subjects who received at least one dose of study drug and had a baseline efficacy measurement
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 142 | 143 | 140
Units on a scale | 1.0 (0.08) | 1.0 (0.14) | 1.0 (0.19)

16. Secondary Outcome: Mean Patient Global Impression of Severity of General Condition Ratings at Day 1
Description: The PGI-S rating scale is the patient's assessment of general condition. The subject rates their overall condition according to the 7 following categories: 1=normal (no sign of illness), 2=borderline ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, and 7=among the most extremely ill. The term "ill" refers to symptoms of jet lag including excessive sleepiness, irritability, malaise, gastrointestinal disturbance, and poor performance. The least squares mean of PGI-S ratings at day 1 is presented here.
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 142 | 143 | 141
units on a scale | 2.2 (0.11) | 1.7 (0.11) | 2.1 (0.11)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.8262, ANOVA
Statistical Analysis 2: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0040, ANOVA

17. Secondary Outcome: Mean Patient Global Impression of Severity of General Condition Ratings at Day 2
Description: The PGI-S rating scale is the patient's assessment of general condition. The subject rates their overall condition according to the 7 following categories: 1=normal (no sign of illness), 2=borderline ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, and 7=among the most extremely ill. The term "ill" refers to symptoms of jet lag including excessive sleepiness, irritability, malaise, gastrointestinal disturbance, and poor performance. The least squares mean of PGI-S ratings at day 2 is presented here.
Time Frame: Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 141 | 142 | 139
units on a scale | 1.6 (0.08) | 1.5 (0.08) | 1.6 (0.08)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.9595, ANOVA
Statistical Analysis 2: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.3539, ANOVA; Least square mean

18. Secondary Outcome: Mean Patient Global Impression of Severity of General Condition Ratings at Day 3
Description: The PGI-S rating scale is the patient's assessment of general condition. The subject rates their overall condition according to the 7 following categories: 1=normal (no sign of illness), 2=borderline ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, and 7=among the most extremely ill. The term "ill" refers to symptoms of jet lag including excessive sleepiness, irritability, malaise, gastrointestinal disturbance, and poor performance. The least squares mean of PGI-S ratings at day 3 is presented here.
Time Frame: Day 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 141 | 141 | 139
units on a scale | 1.2 (0.06) | 1.4 (0.06) | 1.4 (0.06)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.1038, ANOVA
Statistical Analysis 2: Comparison: Armodafinil 150 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.8112, ANOVA

19. Secondary Outcome: Change in State and Trait Anxiety Inventory Total Score From Baseline to Endpoint
Description: The State and Trait Anxiety Inventory is a validated self-reporting instrument used to assess anxiety in adults. The inventory consists of 2 scales, state anxiety, which evaluates how the subject feels currently (transient anxiety), and trait anxiety, which evaluates how the subject feels generally (general tendency towards anxiety). Each scale consists of 20 questions, and a higher score indicates greater anxiety. Scores range from 20 (no anxiety) to 80 (maximum anxiety). The change in total score from Baseline to endpoint is presented here.
Time Frame: Endpoint defined as either Day 3 or last observation after baseline
Population: Safety analysis population defined as all subjects who had at least one dose of study drug and one State and Trait Anxiety Inventory Assessment after Baseline
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 142 | 143 | 141
Units on a scale | 0.0 (5.10) | 1.6 (8.30) | 0.6 (7.0)

20. Secondary Outcome: Change in State and Trait Anxiety Inventory Total Score From Baseline to Day 1
Description: The State and Trait Anxiety Inventory is a validated self-reporting instrument used to assess anxiety in adults. The inventory consists of 2 scales, state anxiety, which evaluates how the subject feels currently (transient anxiety), and trait anxiety, which evaluates how the subject feels generally (general tendency towards anxiety). Each scale consists of 20 questions, and a higher score indicates greater anxiety. Scores range from 20 (no anxiety) to 80 (maximum anxiety). The change in total score from Baseline to Day 1 is presented here.
Time Frame: Day 1
Population: Safety analysis population defined as all subjects who had at least one dose of study drug and completed the State and Trait Anxiety Inventory Assessment at Baseline and Day 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 141 | 140 | 140
Units on a scale | 3.8 (6.8) | 4.3 (8.24) | 4.3 (7.04)

21. Secondary Outcome: Change in State and Trait Anxiety Inventory Total Score From Baseline to Day 2
Description: The State and Trait Anxiety Inventory is a validated self-reporting instrument used to assess anxiety in adults. The inventory consists of 2 scales, state anxiety, which evaluates how the subject feels currently (transient anxiety), and trait anxiety, which evaluates how the subject feels generally (general tendency towards anxiety). Each scale consists of 20 questions, and a higher score indicates greater anxiety. Scores range from 20 (no anxiety) to 80 (maximum anxiety). The change in total score from Baseline to Day 2 is presented here.
Time Frame: Day 2
Population: Safety analysis population defined as all subjects who had at least one dose of study drug and completed the State and Trait Anxiety Inventory Assessment at Baseline and Day 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 139 | 141 | 136
Units on a scale | 1.5 (5.82) | 2.8 (7.52) | 1.3 (6.86)

22. Secondary Outcome: Change in State and Trait Anxiety Inventory Total Score From Baseline to Day 3
Description: The State and Trait Anxiety Inventory is a validated self-reporting instrument used to assess anxiety in adults. The inventory consists of 2 scales: state anxiety, which evaluates how the subject feels currently (transient anxiety), and trait anxiety, which evaluates how the subject feels generally (general tendency towards anxiety). Each scale consists of 20 questions, and a higher score indicates greater anxiety. Scores range from 20 (no anxiety) to 80 (maximum anxiety). The change in total score from Baseline to Day 3 is presented here.
Time Frame: Day 3
Population: Safety analysis population defined as all subjects who had at least one dose of study drug and completed the State and Trait Anxiety Inventory Assessment at Baseline and Day 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 140 | 141 | 138
Units on a scale | -0.1 (5.11) | 1.6 (8.34) | 0.2 (6.6)

23. Secondary Outcome: Mean Change From Baseline to Endpoint in Total Sleep Time as Measured by Nocturnal Polysomnography
Description: Nocturnal Polysomnography records normal and abnormal physiological activity during an entire night's sleep. It documents the adequacy of sleep, including frequency duration, and total amount of stage 1-2, stage 3-4 (slow wave sleep), rapid eye movement sleep, and apnea/hypopnea index. Data presented here represents the difference in mean total sleep time overnight from Baseline to Day 2 as recorded by nocturnal polysomnography.
Time Frame: Baseline and Day 2 (Endpoint)
Population: Safety analysis population defined as all subjects who had at least one dose of study drug and underwent nocturnal polysomnography at Baseline and Day 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 141 | 141 | 138
Minutes | -10.0 (69.76) | -30.5 (83.03) | -5.2 (62.88)

24. Secondary Outcome: Mean Change From Baseline to Endpoint in Latency to Persistent Sleep as Measured by Nocturnal Polysomnography
Description: Nocturnal Polysomnography records normal and abnormal physiological activity during an entire night's sleep. It documents the adequacy of sleep, including frequency duration, and total amount of stage 1-2, stage 3-4 (slow wave sleep), rapid eye movement sleep, and apnea/hypopnea index. Data presented here represents the difference in mean latency to persistent sleep from Baseline to Day 2 as recorded by nocturnal polysomnography.
Time Frame: Baseline and Day 2 (Endpoint)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 141 | 141 | 138
Minutes | -12.9 (36.00) | -0.8 (44.78) | -11.0 (29.56)

25. Secondary Outcome: Mean Change in Sleep Efficiency From Baseline To Endpoint as Measured by Nocturnal Polysomnography
Description: Nocturnal Polysomnography records normal and abnormal physiological activity during an entire night's sleep. It documents the adequacy of sleep, including frequency duration, and total amount of stage 1-2, stage 3-4 (slow wave sleep), rapid eye movement sleep, and apnea/hypopnea index. Data presented here represents the difference in mean sleep efficiency from Baseline to Day 2 as recorded by nocturnal polysomnography. Sleep efficiency is defined as the ratio of time spent asleep (total sleep time) to the amount of time in bed.
Time Frame: Baseline and Day 2 (Endpoint)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 141 | 141 | 138
Percent | -2.1 (14.53) | -6.3 (17.23) | -1.1 (13.10)

26. Secondary Outcome: Mean Change From Baseline to Endpoint in Wake Time After Sleep Onset as Measured by Nocturnal Polysomnography
Description: Nocturnal Polysomnography records normal and abnormal physiological activity during an entire night's sleep. It documents the adequacy of sleep, including frequency duration, and total amount of stage 1-2, stage 3-4 (slow wave sleep), rapid eye movement sleep, and apnea/hypopnea index. Data presented here represents the difference in mean wake time after sleep onset (time spent awake from sleep onset to final awakening) from Baseline to Day 2 as recorded by nocturnal polysomnography.
Time Frame: Baseline and Day 2 (Endpoint)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 141 | 141 | 138
Minutes | 20.0 (70.80) | 30.4 (76.40) | 14.4 (62.18)

ADVERSE EVENTS:
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 0/142 | 0/143 | 0/142
Other Adverse Events (participants affected / at risk) | 44/142 | 67/143 | 41/142
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 50 mg/Day (N=142) | Armodafinil 150 mg/Day (N=143) | Placebo (N=142)
Palpitations (Cardiac disorders) | 1 | 7 | 0
Nausea (Gastrointestinal disorders) | 4 | 18 | 5
Diarrhea (Gastrointestinal disorders) | 6 | 7 | 4
Medical device site reaction (Injury, poisoning and procedural complications) | 23 | 24 | 25
Headache (Nervous system disorders) | 23 | 36 | 16
Dizziness (Nervous system disorders) | 2 | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days